CLINICAL TRIAL: NCT07225803
Title: Management of Dyssynergic Defecation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Adil Bharucha, MBBS, MD, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-003767
Record Dates: First submitted 2025-10-17; First posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Dyssynergic Defecation; Constipation
MeSH Terms: conditions — Constipation | interventions — Biofeedback, Psychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biofeedback and inspiratory muscle training (BFT Plus) (Experimental): Subjects in the BFT Plus arm will participate in a minimum of 6 up to a maximum of 20 biofeedback sessions, with each session lasting approximately 60 minutes.
  In addition, subjects will engage in inspiratory muscle training (IMT) at home.
  Interventions: Behavioral: Biofeedback; Behavioral: Inspiratory muscle training (IMT)
- Biofeedback only (BFT Alone) (Active Comparator): Subjects in the BFT Plus arm will participate in a minimum of 6 up to a maximum of 20 biofeedback sessions, with each session lasting approximately 60 minutes.
  Interventions: Behavioral: Biofeedback

INTERVENTIONS:
Behavioral: Biofeedback — During anorectal biofeedback therapy, subjects are coached to improve abnormal patterns while observing activity recorded by manometry and/or surface EMG (electromyography) on a computer monitor while seated on a chair or a commode.
Behavioral: Inspiratory muscle training (IMT) — Subjects will engage in inspiratory muscle training (IMT) that is tailored to the baseline performance of the individual.
  Arms: Biofeedback and inspiratory muscle training (BFT Plus)

SUMMARY:
The purpose of this research is to better understand constipation and improve biofeedback treatments.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18-80 years who are able and willing to provide written informed consent and to comply with the requirements for the entire study
* Satisfy Rome III criteria for functional constipation and/or irritable bowel syndrome as assessed by questionnaires and objective evidence of dyssynergic defecation on anorectal testing

Exclusion Criteria:

* Clinical evidence of significant cardiovascular, respiratory, renal, hepatic, gastrointestinal, hematological, neurological, psychiatric or other diseases that may interfere with the objectives of the study and/or pose safety concerns.
* History of total, hemi- or subtotal colectomy at any time or other abdominal operations within 60 days prior to entry into the study. Segmental resection of the colon (e.g. sigmoid resection) for diverticulitis will be permitted.
* Current anal fissure
* Clinically significant structural abnormalities (eg, rectocele > 4cm, large enterocele, full thickness rectal prolapse) that, in the opinion of the investigator, are likely contributing to symptoms
* Current or past history of colon or rectal cancer, scleroderma, inflammatory bowel disease, congenital anorectal abnormalities, solitary rectal ulcer syndrome, rectal resection or pelvic irradiation
* Pregnant or nursing women, prisoners and institutionalized individuals
* BMI >35 kg/m2
* Use of opioid analgesics or GLP-1 receptor agonists. Patients on opioids will be allowed to participate if they have discontinued them for at least 1 week before the date of screening and are willing to stay off them for the duration of the study.
* Current use of anticholinergics (eg. amitriptyline, hyoscyamine). Patients who use low dose tricyclic antidepressants (nortriptyline or amitriptyline up to 50 mg/day) will be eligible provided they do not increase the dose during the study period. Patients on higher doses are eligible to participate if it is safe and they are willing to reduce their medication dose at least 3 days (72 hrs) before the date of screening and are willing to stay off them till the study is complete.
* Current use of laxatives (Ex-lax, senna, herbal supplements), linaclotide, lubiprostone, and prucalopride to treat constipation- patients using these medications will be eligible to participate if they can discontinue the medication at least 3 days (72 hrs.) before the date of screening and are willing to stay off them till the study is complete (As detailed later, all participants can use Miralax throughout the study).
* Any other factors that increase the risk to participants of participating in the study and/or undermine the integrity of the data.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-07-18 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Change in rectoanal gradient during evacuation | Baseline, through study completion, an average of 16 weeks
  Rectoanal gradient during evacuation is the pressure difference between the rectum and the anal canal during simulated evacuation, measured in millimeters of mercury (mmHg).
Change in rectal pressure during evacuation | Baseline, through study completion, an average of 16 weeks
  Rectal pressure during evacuation is the difference in rectal pressure during - before evacuation. Results are measured in millimeters of mercury (mmHg).
Change in balloon expulsion time | Baseline, through study completion, an average of 16 weeks
  Rectal balloon expulsion directly assesses evacuation. Patients will be asked to expel a rectal balloon inflated up to 50 ml of water. The time required to expel the balloon will be measured and reported in seconds.
Change in rectal emptying time | Baseline, through study completion, an average of 16 weeks
  Rectal emptying will be assessed via fecoflowmetry by measuring the time required to defecate (seconds) artificial stool from the rectum
Change in rectal emptying rate | Baseline, through study completion, an average of 16 weeks
  Rectal emptying will be assessed via fecoflowmetry by measuring the amount (gm) of artificial stool from the rectum. The 2 metrics - amount and time - are integrated to measure amount (gm) evacuated per unit time (second) (gm/sec).

SECONDARY OUTCOMES:
Change in Patient Assessment of Constipation-Symptoms (PAC-SYM) questionnaire | Baseline, through study completion, an average of 16 weeks, 3 months post completion, 12 months post completion
  The PAC-SYM questionnaire assesses the severity of patient-reported symptoms related to constipation. The questionnaire is divided into three symptom subscales: abdominal (four items); rectal (three items); and stool (five items). Items are scored on 5-point Likert scales, with scores ranging from 0 to 4 (0 = 'symptom absent', 1 = 'mild', 2 = 'moderate', 3 = 'severe' and 4 = 'very severe'). A mean total score in the range of 0-4 is generated by dividing the total score by the number of questions completed; the lower the total score, the lower the symptom burden. Scores range from 0 to 48.
Change in Patient Assessment of Constipation - Quality of Life (PAC-QOL) questionnaire | Baseline, through study completion, an average of 16 weeks, 3 months post completion , 12 months post completion
  The PAC-QOL questionnaire is a patient-reported outcome measure to evaluate quality of life in constipated persons. The questionnaire is divided into four subscales: worries and concerns (11 items), physical discomfort (4 items), psychosocial discomfort (8 items), and satisfaction (5 items). Scale scores represent average item scores and range from 0 to 4, where higher scores represent poorer quality of life. Scores range from 0 to 112.
Physical Activity Rating Scale | Baseline
  Physical Activity Rating is a questionnaire for categorizing physical activity level, which is used in the equation for the non-exercise fitness test. The Physical Activity Rating is a score value between 0 to 7. The non-exercise fitness test of VO2max, a measure of cardiovascular fitness, will be calculated using the following equation:
  56.363 + 1.921 (Physical Activity Rating) - 0.381(Age) - 0.754(Body Mass Index) + 10.987(Sex: 0 for women, 1 for men)
Quebec User Evaluation of Satisfaction with Assistive Technology questionnaire | through study completion, an average of 16 weeks
  Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST) 11-item questionnaire is a standardized tool to measure the satisfaction of an individual who is using an assistive device. It inquiries about the assistive device itself: dimensions, weight, ease of adjustment, safety, durability, ease of use, comfortability, and effectiveness; and service: service delivery, maintenance, professional services, and follow up services. Each question is answered on a Likert scale, where 1 = not satisfied at all, and 5 = very satisfied. Possible scores range from 11 to 55.
Change in stool frequency | Baseline, through study completion, an average of 16 weeks, 3 months post completion, 12 months post completion
  Daily number of bowel movements will be self-reported by participants via a bowel diary.
Change in stool consistency | Baseline, through study completion, an average of 16 weeks, 3 months post completion, 12 months post completion
  Daily stool consistency will be self-reported by participants via a bowel diary by using the Bristol Stool Chart. Participants will compare stool's appearance to the 7 types and selecting the one that most closely matches. Type 1-2 indicate constipation, Type 3-4 are ideal stools as they are easier to pass, and Type 5-7 may indicate diarrhea and urgency.
Change in anal digitation | Baseline, through study completion, an average of 16 weeks, 3 months post completion, 12 months post completion
  The total number of times anal digitation was required to achieve a bowel movement will be self-reported via the bowel diary.
Change in sense of incomplete evacuation | Baseline, through study completion, an average of 16 weeks, 3 months post completion, 12 months post completion
  The total number of times a participant felt a sense of incomplete evacuation after a bowel movement will be self-reported via the bowel diary.
Change in spontaneous bowel movements | Baseline, through study completion, an average of 16 weeks, 3 months post completion, 12 months post completion
  The total number of times a participant achieves a spontaneous bowel movement will be self-reported via the bowel diary.
Change in pain during bowel movements | Baseline, through study completion, an average of 16 weeks, 3 months post completion, 12 months post completion
  Pain during bowel movements will be self-reported by participants via the bowel diary using a 4-point Likert scale (0 = None, 1 = Mild, 3 = Moderate, and 4 = Severe).
Change in bowel symptoms before and after biofeedback therapy | Baseline, through study completion, an average of 16 weeks, 3 months post completion, 12 months post completion
  Bowel symptoms pre and post biofeedback therapy will be assessed using a self-reported questionnaire. The survey includes Severity of constipation, satisfaction with bowel movements, satisfaction with current treatment of constipation, severity of constipation compared to baseline, adequate relief of constipation, use of laxatives, and severity of abdominal bloating and distention. Impact of constipation on 15 QOL domains.
Change in Hospital Anxiety and Depression (HAD) score | Baseline, through study completion, an average of 16 weeks
  The Hospital Anxiety and Depression (HAD) is a self-reported 14 item questionnaire asking participants to reflect on their mood in the past week. . Each item is rated on a 4-point scale, for a total score ranging from 0-21 for each subscale. A higher score indicates higher distress.
Change in forced vital capacity | Baseline, through study completion, an average of 16 weeks
  Forced vital capacity (FVC) is the the total volume of air exhaled with maximal effort, and is measured using a spirometer (reported in liters).
Change in forced expiratory volume | Baseline, through study completion, an average of 16 weeks
  Forced expiratory volume (FEV) is the total volume of air exhaled with maximal effort, and is measured using a spirometer (reported in liters).
Change in forced expiratory time | Baseline, through study completion, an average of 16 weeks
  Forced expiratory time (FET) is the time taken to exhale the greatest volume of air from the lungs as possible and is measured using a spirometer (reported in seconds).
Change in peak inspiratory flows | Baseline, through study completion, an average of 16 weeks
  Peak inspiratory flow (PIF) is the maximum volume and rate of air that can be forcefully inhaled out of the lungs, and is measured using a spirometer (reported in liters per second (L/sec)).
Change in peak expiratory flows | Baseline, through study completion, an average of 16 weeks
  Peak expiratory flow (PEF) is the maximum volume and rate of air that can be forcefully exhaled out of the lungs and is measured using a spirometer (reported in in liters per second (L/sec)).
Change in forced expiratory volume/forced vital capacity ratio | Baseline, through study completion, an average of 16 weeks
  The total volume of air exhaled with maximal effort / The volume of air exhaled with maximum effort in the first second (reported as percentage).
Change in forced expiratory flow at 25-75% of forced vital capacity | Baseline, through study completion, an average of 16 weeks
  The average flow from the point at which 25% of the forced vital capacity has been exhaled to the point at which 75% of the forced vital capacity has been exhaled. A reduced forced expiratory flow 25-75% is a marker of small airway obstruction.
Change in forced expiratory flow at 50% of forced vital capacity | Baseline, through study completion, an average of 16 weeks
  The flow rate at the point at which 50% point of the forced vital capacity has been exhaled, and is a marker of small airway obstruction.
Change in forced inspiratory vital capacity | Baseline, through study completion, an average of 16 weeks
  Forced inspiratory vital capacity is the maximum volume of air that can be inhaled after a full expiration (reported in liters).
Change in peak inspiratory pressure | Baseline, through study completion, an average of 16 weeks
  Peak inspiratory pressure is the peak pressure during forceful inspiration against an occluded airway (Mueller maneuver), reported in liters per minute (L/min)
Change in peak expiratory pressure | Baseline, through study completion, an average of 16 weeks
  Peak expiratory pressure is the peak pressure during forceful expiration against an occluded airway (Valsalva maneuver), reported in liters per minute (L/min)

CONTACTS AND LOCATIONS:
Overall Officials: Adil E. Bharucha, MBBS, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials/cls-20450326